CLINICAL TRIAL: NCT01710202
Title: Sensitivity of Short and Long Allele Carriers of the 5-HTTLPR to Environmental Threat Post Hydrocortisone Administration
Acronym: 5-HTTLPR
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-12-0017
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder; Anxiety Disorders
Keywords: Hydrocortisone; Cortisol; Testosterone; Stress; Serotonin; 5-HTTLPR; Amygdala; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Depression | interventions — Hydrocortisone

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Placebo: Control group who will not receive hydrocortisone. Will act as a comparison group to the hydrocortisone group.
- Experimental: Hydrocortisone: Group will receive 20mg oral hydrocortisone
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Each subject in this group will receive one 20mg hydrocortisone capsule to be taken by mouth.
  Other Names: Cortef; Cortisol; Hydrocortone
  Groups: Experimental: Hydrocortisone

SUMMARY:
The current study will test the causal relationship between elevated levels of cortisol and the serotonin transporter gene (5-HTTLPR) as these factors influence sensitivity to environmental threat. The investigators predict that carriers of the short allele of the serotonin transporter gene who have elevated cortisol levels will be most sensitive to threatening environments, whereas carriers of the long allele who do not have elevated cortisol (placebo subjects) will be least sensitive.

DETAILED DESCRIPTION:
Depression vulnerability has been linked to certain variants of the serotonin transporter gene. Research indicates that a polymorphism of the serotonin transporter (5-HTTLPR) gene appears to moderate the association between life stress and depression onset. Life stress robustly predicts depression onset for individuals with two short 5-HTTLPR alleles. Individuals homozygous for the short 5-HTTLPR allele thus appear to be more sensitive to the effect of life stress, which in turn contributes to depression onset. A recent study showed that short allele carriers presented with a threat (social or other threats) who also had high levels of testosterone had elevated cortisol after exposure to the threat. There is neurobiological evidence that short allele status, elevated testosterone levels, and elevated cortisol levels are all linked to amygdala hyper-reactivity to the same classes of environmental threats. Thus, this study will test, for the first time, a potential interaction between 5-HTTLPR status and experimentally manipulated cortisol levels as risk factors for downstream mood and/or anxiety disorders by examining potential dysregulated stress responses among short allele carriers who have elevated cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* Are you under the age of 18 years old?
* Have you ever had an allergic reaction to hydrocortisone?
* Do you have diabetes or high blood pressure?
* Do you have any thyroid, liver, heart, lung, or kidney problems?
* Do you have herpes, HIV or any sexual transmitted disease?
* Are you currently pregnant or think you might be pregnant? Have you taken RU486, Plan B or "Morning After Pill" within the last 2 weeks? - Are you currently breastfeeding?
* Have you been sick within the last week? Do you have any fungal infections?
* Have you been exposed to measles or chicken pox in the last week?
* Have you ever had a seizure?
* Do you have any disease of bony tissue, such as osteoporosis?
* Do you have any autoimmune diseases, such as myasthenia gravis?
* Do you have multiple sclerosis?
* Do you have any condition that compromises you immune system function or causes you to be more likely to get sick?
* Have you had any recent surgeries?
* Do you have and gastrointestinal problems, such as ulcers, diverticulitis, colitis, hepatitis, or Crohn disease?
* Are you taking any of the following medications: nevirapine, telbivudine, sipuleucel-T (IV), natalizumab (IV)?
* Have you received any vaccinations within the last week?
* With the exception of vitamins, have you taken any medications in the last 3 days, including all over-the counter medications and/or supplements (e,g. Tylenol, ibuprofen, St. John's Wort, cold remedies)?
* Do you currently have or have you had in the past of any kind of cancer?
* Do you have any significant medical or psychiatric illnesses not listed above?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Texas at Austin students
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in testosterone concentration | 2 hours post hydrocortisone administration
  Subjects will be administered hydrocortisone or placebo. One hour after administration, they will be exposed to an environmental threat manipulation. 20 minutes after this manipulation, saliva will be collected, and testosterone concentrations will be assessed and compared to pre-manipulation concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, Ph.D., Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - University of Texas at Austin Department of Psychology, Austin, Texas
  - University of Texas at Austin, Austin, Texas

REFERENCES:
- [Background] Josephs RA, Telch MJ, Hixon JG, Evans JJ, Lee H, Knopik VS, McGeary JE, Hariri AR, Beevers CG. Genetic and hormonal sensitivity to threat: testing a serotonin transporter genotype x testosterone interaction. Psychoneuroendocrinology. 2012 Jun;37(6):752-61. doi: 10.1016/j.psyneuen.2011.09.006. Epub 2011 Oct 5. PMID 21978869